CLINICAL TRIAL: NCT00686023
Title: Comparing Surgical Techniques for CRIF of Pertrochanteric Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: MD Eli Steinberg, orthopedic trauma manager department B, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-08-ES-0054
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Femur Fracture
Keywords: pertrochanteric femur fracture; DHS; IMN
MeSH Terms: conditions — Femoral Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): DHS fixation
  Interventions: Procedure: internal fixation (DHS - richard nail)
- 2 (Active Comparator): IMN fixation
  Interventions: Procedure: internal fixation (inflatable PFN by DISCOTEC)

INTERVENTIONS:
Procedure: internal fixation (DHS - richard nail) — internal fixation
  Other Names: DHS - richard nail
  Arms: 1
Procedure: internal fixation (inflatable PFN by DISCOTEC) — internal fixation
  Other Names: inflatable PFN by DISCOTEC
  Arms: 2

SUMMARY:
Hypothesis: Inflatable intra medullary femoral nailing is superior to DHS in terms of blood loss, operative complications and postoperative rehabilitation in the management of pertrochanteric femur neck fractures.

DETAILED DESCRIPTION:
patients with pertrochanteric fractures of the femur will be randomly assigned to one of 2 groups.

group 1 will undergo internal fixation using a DHS device. group 2 will undergo internal fixation using an inflatable intramedullary femoral nail device post operative care will be the same including DVT prophylaxis, early mobilization.

weight baring will be aloud in cases of a stable fracture (EVANS 1-3) non weight bearing until callus bridge in patients with unstable fractures (EVANS 4-6)

outcomes: death within first year

postoperative complications length of hospitalization time to mobilization functional score reontgenic evaluation

ELIGIBILITY:
Inclusion Criteria:

* Pertrochanteric femur fracture
* Unilateral
* Age over 60 years
* Low energy trauma
* ASA score 0-3

Exclusion Criteria:

* Reverse oblique fractures
* Pathological fractures
* Severe osteoarthritis of the hip joint
* Previous operations on same leg
* ASA score 4-5

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
death within 1 year of operation | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Eli Steinberg, MD, Principal Investigator — TASMC
Locations (1):
- TASMC, Tel Aviv, Israel

REFERENCES:
- [Result] Folman Y, Ron N, Shabat S, Hopp M, Steinberg E. Peritrochanteric fractures treated with the Fixion expandable proximal femoral nail: technical note and report of early results. Arch Orthop Trauma Surg. 2006 Apr;126(3):211-4. doi: 10.1007/s00402-006-0110-0. Epub 2006 Feb 24. PMID 16501984
- [Result] Lepore L, Lepore S, Maffulli N. Intramedullary nailing of the femur with an inflatable self-locking nail: comparison with locked nailing. J Orthop Sci. 2003;8(6):796-801. doi: 10.1007/s00776-003-0709-8. PMID 14648267
- [Result] Pajarinen J, Lindahl J, Michelsson O, Savolainen V, Hirvensalo E. Pertrochanteric femoral fractures treated with a dynamic hip screw or a proximal femoral nail. A randomised study comparing post-operative rehabilitation. J Bone Joint Surg Br. 2005 Jan;87(1):76-81. PMID 15686241
- [Result] Leung KS, So WS, Shen WY, Hui PW. Gamma nails and dynamic hip screws for peritrochanteric fractures. A randomised prospective study in elderly patients. J Bone Joint Surg Br. 1992 May;74(3):345-51. doi: 10.1302/0301-620X.74B3.1587874.
- [Result] Hardy DC, Descamps PY, Krallis P, Fabeck L, Smets P, Bertens CL, Delince PE. Use of an intramedullary hip-screw compared with a compression hip-screw with a plate for intertrochanteric femoral fractures. A prospective, randomized study of one hundred patients. J Bone Joint Surg Am. 1998 May;80(5):618-30. doi: 10.2106/00004623-199805000-00002. PMID 9611022